CLINICAL TRIAL: NCT06113419
Title: Timing of CHolecystectomy In Severe PAncreatitis (CHISPA): Study Protocol for a Randomized Controlled Trial.
Brief Title: Timing of CHolecystectomy In Severe PAncreatitis
Acronym: CHISPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Mayor Méderi (Other)
Collaborators: Universidad del Rosario (Other)
Responsible Party: Principal Investigator, Camilo Ramirez Giraldo, General Surgeon, Hospital Universitario Mayor Méderi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-26-02B; DVO005 2456-CV1683 (Other: Universidad del Rosario's Ethics Committee)
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Acute Pancreatitis; Cholelithiasis
Keywords: cholecystectomy; Acute Pancreatitis; Cholelithiasis
MeSH Terms: conditions — Pancreatitis; Cholelithiasis | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Intervention Model Description: CHISPA is a randomized controlled, parallel-group, superiority clinical trial. Patients will be randomly allocated to receive early laparoscopic cholecystectomy (within 72 hours after randomization) or interval laparoscopic cholecystectomy (30 +/- 5 days after randomization).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early cholecystectomy (Experimental): Early laparoscopic cholecystectomy (within 72 hours after randomization)
  Interventions: Procedure: Laparoscopic cholecystectomy
- Interval cholecystectomy (Active Comparator): Interval laparoscopic cholecystectomy (30 +/- 5 days after randomization).
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — Laparoscopic cholecystectomy will be performed using the standard American 4-port technique, insufflation will be achieved using CO2 to 15mmHg of pressure. Calot's triangle will be dissected until the critical view of safety is reached, being careful to dissect above the R4U line. After reaching the critical view of safety, two proximal and one distal clip will be placed on both the cystic conduct and artery separately, cutting the clips and then dissecting the gallbladder in a cystfundic direction. When the critical view of safety is not reached, the surgeon may perform a fundus-first cholecystectomy, subtotal cholecystectomy, conversion to open procedure, intraoperative cholangiography or cholecystostomy to their own discretion. It will also be the surgeon's criteria to employ or not a drain system in the surgical site. The decision for theses interventions will be taken intraoperatively and will be according to findings during the procedure.

SUMMARY:
The goal of this clinical trial is to compare outcomes for interval or early laparoscopic cholecystectomy in patients with moderately severe and severe pancreatitis. The main question[s] it aims to answer are:

* To establish whether there is a difference in surgical outcomes comparing patients diagnosed with severe or moderately severe pancreatitis on which early cholecystectomy was performed versus performing interval cholecystectomy.
* The primary endpoint will be to evaluate major complications, defined as a Clavien-Dindo score greater than or equal to III/V.
* Secondary endpoints include evaluating minor complications (defined as a Clavien-Dindo score below III/V), biliary disease recurrence, mortality, postoperative hospital stay and postoperative admittance into an intensive care unit.

Participants will be randomly assigned to either group: early cholecystectomy during the pancreatitis hospitalization or interval cholecystectomy scheduled 4 weeks after clinical resolution of pancreatitis.

DETAILED DESCRIPTION:
CHISPA is a randomized controlled, parallel-group, superiority clinical trial. An intention- to-treat analysis will be performed. It seeks to evaluate differences between patients taken to early cholecystectomy during hospital admission (72 hours after randomization) versus delayed cholecystectomy (30 +/- 5 days after randomization). Primary endpoint is major complications associated to laparoscopic cholecystectomy defined as a Clavien-Dindo score of over III/V during the first 90 days after the procedure. Secondary endpoints include recurrence of biliary disease, mortality, minor complications (Clavien-Dindo score below III/V), days of postoperative hospital stay, and days admitted in an intensive care unit postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, diagnosis of pancreatitis according to Atlanta guidelines, moderately severe or severe pancreatitis (APACHE score ≥8 on admittance)
* Biliary pancreatitis diagnosed on imaging (be it ultrasound, magnetic resonance imaging and/or tomography)
* Recovery of pancreatitis by tolerance of oral intake (defined as 24 hours of food consumption of any consistency without emetic episodes and pain defined as 4/10 on the visual analogue score of pain) and written informed consent.

Exclusion Criteria:

* Pregnancy
* History of cholecystectomy
* Planned open cholecystectomy
* Pancreatitis-associated complication before laparoscopic cholecystectomy (compartment syndrome, bleeding and/or need for peripancreatic collection drainage)
* Chronic pancreatitis,
* More than one episode of pancreatitis
* Active malignant disease
* Septic shock
* Choledocholithiasis not resolved by ERCP, post-ERCP perforation and post-ERCP concomitant pancreatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Major complications (rates) | 90 days
  Clavien-Dindo score III in patients with moderately severe and severe acute pancreatitis of biliary origin taken to early vs interval cholecystectomy
Major complications (rates) | 90 days
  Clavien-Dindo score IV in patients with moderately severe and severe acute pancreatitis of biliary origin taken to early vs interval cholecystectomy
Major complications (rates) | 90 days
  Clavien-Dindo score V in patients with moderately severe and severe acute pancreatitis of biliary origin taken to early vs interval cholecystectomy

SECONDARY OUTCOMES:
Recurrence (rates) | 90 days
  Biliary disease recurrence defined as a new admission for recurrent pancreatitis, cholecystitis, cholangitis, choledocholithiasis, need fro ERCP or biliary colic previous to the surgical procedure until 90 postoperative days after it
Mortality (rates) | 90 days
  Determine differences in mortality between patients with moderately severe and severe acute pancreatitis of biliary origin taken to early vs interval cholecystectomy
Postoperative hospital stay length (days; median) | 90 days
  Compare differences in postoperative hospital stay length (general) in patients with moderately severe and severe acute pancreatitis of biliary origin taken to early vs interval cholecystectomy
Minor complications (rates) | 90 days
  Clavien-Dindo score I-II in patients with moderately severe and severe acute pancreatitis of biliary origin taken to early vs interval cholecystectomy
Postoperative stay length in the ICU (days; median) | 90 days
  Compare differences in postoperative stay length in the ICU in patients with moderately severe and severe acute pancreatitis of biliary origin taken to early vs interval cholecystectomy

CONTACTS AND LOCATIONS:
Overall Officials: Camilo Ramirez-Giraldo, MD, Principal Investigator — Hospital Universitario Mayor Méderi
Locations (2):
- Colombia (2):
  - Hospital Universitario Mayor-Méderi, Bogota, Cundinamarca
  - Hospital Universitario Méderi Barrios Unidos, Bogota, Cundinamarca

IPD SHARING:
Plan to Share IPD: Yes
Data obtained and input into the database is anonymous, without any individual or identifying characteristics will be stored in a dataset from the Centro de Recursos para el Aprendizaje y la Investigación, property of and administered by the Universidad del Rosario as a plan of data management. Moreover, the different codes used in the analysis will be stored in this dataset.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: It is in our plans once we obtain a register number from Clinical Trials in order to publish the protocol, statistical analysis plan and clinical study report in a scientific journal so it will be available to all people interested.
Access Criteria: It is in our plans to be published in a scientific journal available to all people interested.

REFERENCES:
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Background] Yokoe M, Takada T, Mayumi T, Yoshida M, Isaji S, Wada K, Itoi T, Sata N, Gabata T, Igarashi H, Kataoka K, Hirota M, Kadoya M, Kitamura N, Kimura Y, Kiriyama S, Shirai K, Hattori T, Takeda K, Takeyama Y, Hirota M, Sekimoto M, Shikata S, Arata S, Hirata K. Japanese guidelines for the management of acute pancreatitis: Japanese Guidelines 2015. J Hepatobiliary Pancreat Sci. 2015 Jun;22(6):405-32. doi: 10.1002/jhbp.259. Epub 2015 May 13. PMID 25973947
- [Background] Leppaniemi A, Tolonen M, Tarasconi A, Segovia-Lohse H, Gamberini E, Kirkpatrick AW, Ball CG, Parry N, Sartelli M, Wolbrink D, van Goor H, Baiocchi G, Ansaloni L, Biffl W, Coccolini F, Di Saverio S, Kluger Y, Moore E, Catena F. 2019 WSES guidelines for the management of severe acute pancreatitis. World J Emerg Surg. 2019 Jun 13;14:27. doi: 10.1186/s13017-019-0247-0. eCollection 2019. PMID 31210778
- [Background] Prasanth J, Prasad M, Mahapatra SJ, Krishna A, Prakash O, Garg PK, Bansal VK. Early Versus Delayed Cholecystectomy for Acute Biliary Pancreatitis: A Systematic Review and Meta-Analysis. World J Surg. 2022 Jun;46(6):1359-1375. doi: 10.1007/s00268-022-06501-4. Epub 2022 Mar 19. PMID 35306590
- [Background] Forsmark CE, Vege SS, Wilcox CM. Acute Pancreatitis. N Engl J Med. 2016 Nov 17;375(20):1972-1981. doi: 10.1056/NEJMra1505202. No abstract available. PMID 27959604
- [Background] Nealon WH, Bawduniak J, Walser EM. Appropriate timing of cholecystectomy in patients who present with moderate to severe gallstone-associated acute pancreatitis with peripancreatic fluid collections. Ann Surg. 2004 Jun;239(6):741-9; discussion 749-51. doi: 10.1097/01.sla.0000128688.97556.94. PMID 15166953
- [Background] Ackermann TG, Cashin PA, Alwan M, Wewelwala CC, Tan D, Vu AN, Bowers KA, Berry R, Croagh DG. The Role of Laparoscopic Cholecystectomy After Severe and/or Necrotic Pancreatitis in the Setting of Modern Minimally Invasive Management of Pancreatic Necrosis. Pancreas. 2020 Aug;49(7):935-940. doi: 10.1097/MPA.0000000000001601. PMID 32658078
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Gupta V, Jain G. Safe laparoscopic cholecystectomy: Adoption of universal culture of safety in cholecystectomy. World J Gastrointest Surg. 2019 Feb 27;11(2):62-84. doi: 10.4240/wjgs.v11.i2.62. PMID 30842813
- [Background] Working Group IAP/APA Acute Pancreatitis Guidelines. IAP/APA evidence-based guidelines for the management of acute pancreatitis. Pancreatology. 2013 Jul-Aug;13(4 Suppl 2):e1-15. doi: 10.1016/j.pan.2013.07.063. PMID 24054878
- [Background] Tenner S, Baillie J, DeWitt J, Vege SS; American College of Gastroenterology. American College of Gastroenterology guideline: management of acute pancreatitis. Am J Gastroenterol. 2013 Sep;108(9):1400-15; 1416. doi: 10.1038/ajg.2013.218. Epub 2013 Jul 30. PMID 23896955
- [Background] Li J, Chen J, Tang W. The consensus of integrative diagnosis and treatment of acute pancreatitis-2017. J Evid Based Med. 2019 Feb;12(1):76-88. doi: 10.1111/jebm.12342. PMID 30806495
- [Background] Sun W, An LY, Bao XD, Qi YX, Yang T, Li R, Zheng SY, Sun DL. Consensus and controversy among severe pancreatitis surgery guidelines: a guideline evaluation based on the Appraisal of Guidelines for Research and Evaluation II (AGREE II) tool. Gland Surg. 2020 Oct;9(5):1551-1563. doi: 10.21037/gs-20-444. PMID 33224831
- [Background] Hughes DL, Morris-Stiff G. Determining the optimal time interval for cholecystectomy in moderate to severe gallstone pancreatitis: A systematic review of published evidence. Int J Surg. 2020 Dec;84:171-179. doi: 10.1016/j.ijsu.2020.11.016. Epub 2020 Nov 20. PMID 33227531
- [Background] da Costa DW, Bouwense SA, Schepers NJ, Besselink MG, van Santvoort HC, van Brunschot S, Bakker OJ, Bollen TL, Dejong CH, van Goor H, Boermeester MA, Bruno MJ, van Eijck CH, Timmer R, Weusten BL, Consten EC, Brink MA, Spanier BWM, Bilgen EJS, Nieuwenhuijs VB, Hofker HS, Rosman C, Voorburg AM, Bosscha K, van Duijvendijk P, Gerritsen JJ, Heisterkamp J, de Hingh IH, Witteman BJ, Kruyt PM, Scheepers JJ, Molenaar IQ, Schaapherder AF, Manusama ER, van der Waaij LA, van Unen J, Dijkgraaf MG, van Ramshorst B, Gooszen HG, Boerma D; Dutch Pancreatitis Study Group. Same-admission versus interval cholecystectomy for mild gallstone pancreatitis (PONCHO): a multicentre randomised controlled trial. Lancet. 2015 Sep 26;386(10000):1261-1268. doi: 10.1016/S0140-6736(15)00274-3. PMID 26460661
- [Background] Sinha R. Early laparoscopic cholecystectomy in acute biliary pancreatitis: the optimal choice? HPB (Oxford). 2008;10(5):332-5. doi: 10.1080/13651820802247078. PMID 18982148
- [Derived] Ramirez-Giraldo C, Conde Monroy D, Daza Vergara JA, Isaza-Restrepo A, Van-Londono I, Trujillo-Guerrero L. Timing of CHolecystectomy In Severe PAncreatitis (CHISPA): study protocol for a randomized controlled trial. BMJ Surg Interv Health Technol. 2024 Mar 7;6(1):e000246. doi: 10.1136/bmjsit-2023-000246. eCollection 2024. PMID 38463464